CLINICAL TRIAL: NCT03583983
Title: Evaluating the Impact of Personalized Recommendations on Healthy Behaviours and Cardio-metabolic Risk
Brief Title: The DNA-Based Lifestyle Enhancement Trial
Acronym: DNAble
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: GeneBlueprint Corp (Unknown); Federal Economic Development Agency for Southern Ontario (FedDev Ontario) (Other); GoodLife Fitness (Unknown); Southlake Regional Health Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20170928
Record Dates: First submitted 2018-06-13; First posted 2018-07-12 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Health Behavior; Genetic Information; Cardiovascular Risk Factor
Keywords: Physical Activity; Dietary Habits; Genetic Scores; Cardiovascular Health
MeSH Terms: conditions — Health Behavior; Motor Activity; Feeding Behavior

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants will be randomized to intervention or control groups using a minimization scheme which will adaptively weight probabilities of treatment assignment based on the distribution of age (> 40 vs. < 40), gender (male vs. female), and ethnicity (European/African/East Asian/South Asian/Latino/Other). This design has been adopted to minimize unintended covariate biases, which can plague smaller trials. Randomization will be implemented through a centralized database. The intervention will be delivered via automated e-mails, minimizing direct personal contact with the intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized Health Recommendations (Other)
  Interventions: Behavioral: Personalized Health Recommendations
- No Health Recommendations (Other)
  Interventions: Behavioral: Generic Health Recommendations

INTERVENTIONS:
Behavioral: Personalized Health Recommendations — Includes 3-month gym membership, personalized exercise and meal plans, and genetic information related to health and wellness traits. The genetic information provided to study participants will consist of scores ranging from 0 to 100 based on the population percentile of the combined effects of many genetic variants, herein referred to as polygenic scores (PGS). PGS for approximately twenty traits related to health, fitness and nutrition will be provided to study participants. These traits are chosen for their relevance to healthy lifestyle habits (e.g. genetic predisposition to adiposity or muscle strength), entertainment value (e.g. preference for mornings) or both (e.g. bitterness taste perception, which while entertaining can also help guide vegetable choices).
  Arms: Personalized Health Recommendations
Behavioral: Generic Health Recommendations — Includes 3-month gym membership and generic recommendations (Canada Food Guide / Health Canada Physical Activity guidelines)
  Arms: No Health Recommendations

SUMMARY:
Despite the known cardiovascular benefits of regular physical activity and having a balanced diet, it has proven challenging to change health behaviours towards favourable lifestyles. The overarching aim of the study is to test the effect of providing personalized genetic information along with diet and exercise plans on adherence to healthy lifestyle habits and cardio-metabolic risk. There is tremendous public interest in genetics and some evidence that providing genetic information can help improve health habits. However, no intervention to date has examined the effect of comprehensive genetic testing using cutting-edge polygenic score (PGS) prediction and an interactive health portal on health behaviours and cardio-metabolic risk. The investigators hypothesize that providing participants with detailed genetic information about genetic determinants of fitness and nutrition traits will help motivate people to adopt healthy lifestyle habits. The primary objective is to test the effect of providing genetic information and interactive recommendations for diet and exercise on adoption of healthy behaviours. The secondary objective is to evaluate the effects of the personalized health recommendations on cardio-metabolic risk markers, such as dyslipidemia, inflammatory markers, and fasting glucose.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is a leading cause of death and disability worldwide, accounting for 17.9 million deaths and the loss of 348 million disability-adjusted life years in 2015 alone. Diabetes and obesity are very strong risk factors for CVD. Individuals with diabetes and obesity have an 82.75% life-time risk for developing CVD. While treatments do exist for both obesity (e.g. bariatric surgery) and diabetes (e.g. pharmaceutical control of blood sugar levels), these only partially attenuate risk of adverse health outcomes and they do not address prevention and upstream causes of cardiovascular diseases, namely sedentary lifestyle and unhealthy diet. Despite the known cardiovascular benefits of regular physical activity and having a balanced diet, it has proven challenging to change health behaviours towards favourable lifestyles. Indeed, the prevalence of obesity is increasing in Canada as less than 80% of adults follow the current recommendation of 150 minutes of moderate-to-vigorous physical activity per week and approximately less than 60% of adults consume fruits and vegetables 5 or more times a day. The overarching aim of the study is to test the effect of providing personalized genetic information along with diet and exercise plans on adherence to healthy lifestyle habits and cardio-metabolic risk. There is tremendous public interest in genetics and some evidence that providing genetic information can help improve health habits. However, no intervention to date has examined the effect of comprehensive genetic testing using cutting-edge polygenic score (PGS) prediction and an interactive health portal on health behaviours and cardio-metabolic risk.

The investigators hypothesize that providing participants with detailed genetic information about genetic determinants of fitness and nutrition traits will help to motivate people to adopt healthy lifestyle habits. The primary objective is to test the effect of providing genetic information and interactive recommendations for diet and exercise on adoption of healthy behaviours. The secondary objective is to evaluate the effects of the personalized health recommendations on cardio-metabolic risk markers, such as dyslipidemia, inflammatory markers, and fasting glucose.

The investigators propose to conduct a randomized controlled trial investigating whether personalized lifestyle recommendations including genetic information motivates Hamilton Health Sciences employees to adopt healthy lifestyle changes. Study participation will be open to Hamilton Health Sciences employees. Recruitment will begin in March 2017. Eligible and consenting individuals will be enrolled. Enrollment will occur in a staggered fashion. The intervention group will receive (1) a free 3-month GoodLife Fitness gym membership providing access to any Ontario GoodLife Fitness facility, (2) professional trainer-approved workout plans, (3) dietitian-approved meal plans, and (4) genetic information pertaining to their health and fitness. The control group will also receive a GoodLife Fitness membership to ensure that all study participants are granted similar ease-of-access to perform physical activities and generic health recommendations (Canadian Food Guide / Health Canada Physical Activity Recommendations) but will not receive the personalized component of the intervention (workout plans, meal plans or genetic information) until the end of their trial period. Participants will be randomized to treatment or control groups using a minimization scheme for adaptive randomization, which will serve to balance age, gender, and ethnicity across groups as participants are enrolled. Thus, randomization will be performed in a single-blind fashion wherein the study team is unaware of whom is receiving the intervention or control. All study participants will be monitored over the course of 3 months beginning with their baseline assessment and ending with their 3-month follow-up assessment. At these two timepoints, study participants will be assessed for behavioural (physical activity levels and diet healthiness), fitness markers (blood pressure, resting heart rate, body fat %, and other anthropometric measurements) and biological markers (lipids, insulin sensitivity, and inflammation) of cardio-metabolic disease.

ELIGIBILITY:
Inclusion Criteria:

* Hamilton Health Science employees living in Southern Ontario who are capable and willing to follow an exercise and diet program for 3 months as well as fitness and blood assessments

Exclusion Criteria:

* Insulin-dependent diabetes
* History of cardiovascular disease (stroke, heart attack, coronary artery bypass graft (CABG) surgery, coronary angioplasty, peripheral artery disease)
* Injury or condition impeding ability to engage in physical activity (e.g. osteoarthritis, COPD)
* Pregnant or breast-feeding or planning to be pregnant
* Anyone on medication that interacts with foods
* Anyone planning to be on vacation for > 2 weeks in the next 3 months.
* Dietary restrictions (e.g. vegetarianism, gluten sensitivity, etc.)
* History of bone marrow transplant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 424 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-01-03 (Actual)

PRIMARY OUTCOMES:
Change in Physical Activity Levels (Strength Training) | Baseline and 3 months follow-up
  Physical activity levels (strength training) will be defined by frequency of strength training per week. Strength training is one of the domains of physical activity recognized by the Canadian Physical Activity Guidelines, which recommend at least two sessions of strength training per week. Accordingly, physical activity levels will be ascertained through the following survey question: "In the last 3 months, how many times per week did you perform strength training?" The minimum value for this outcome would be 0 and there is no theoretical maximum though we expect most values to be below 7 since 7 would represent strength training on a daily basis. Higher values indicate higher levels of physical activity and vice versa.
Change in Physical Activity Levels (Aerobic Exercise) | Baseline and 3 months follow-up
  Physical activity levels (aerobic exercise) will be defined by frequency of aerobic exercise per week. Aerobic exercise is one of the domains of physical activity recognized by the Canadian Physical Activity Guidelines, which recommend at least 150 minutes of moderate to vigorous physical activity per week. Accordingly, physical activity levels will be ascertained through the following survey question: "In the last 3 months, how many times per week did you perform aerobic exercises training?" The minimum value for this outcome would be 0 and there is no theoretical maximum though we expect most values to be below 7 since 7 would represent aerobic exercise on a daily basis. Higher values indicate higher levels of physical activity and vice versa.
Change in Dietary Healthiness | Baseline and 3 months follow-up
  Dietary healthiness will be ascertained using the dietary risk score developed by the INTERHEART study which was found to explain 30% of the population attributable risk for acute myocardial infarction. Briefly, the dietary risk score takes into account consumption of meat, salty snacks, fried foods, fruits and vegetables. The point score ranges from 0 to 6 with higher scores indicating a less healthy diet.

SECONDARY OUTCOMES:
Change in Triglycerides | Baseline and 3 months follow-up
  Serum Triglyceride Levels (mmol/L)
Change in C-Reactive Protein | Baseline and 3 months follow-up
  High Sensitivity Serum C-reactive protein Levels (mg/L)
Change in Fasting Glucose | Baseline and 3 months follow-up
  Serum Fasting Glucose Levels (mmol/L)
Change in Blood Pressure | Baseline and 3 months follow-up
  Blood Pressure (mmHg). Both systolic and diastolic blood pressures will be assessed.
Change in Resting Heart Rate | Baseline and 3 months follow-up
  Resting Heart Rate (Beats / min)
Change in Body Fat % | Baseline and 3 months follow-up
  Body Fat (%)
Change in Circumference of Body Parts | Baseline and 3 months follow-up
  Circumference of thigh, calf, bicep, and shoulder span (millimeters)
Change in Body Mass Index | Baseline and 3 months follow-up
  Body Mass Index - derived from height and weight (weight in kg / height in m ^2)
Change in Cardio-metabolic Risk Score | Baseline and 3 months follow-up
  Cardio-metabolic risk estimated by the validated INTERHEART modified risk score. This score was developed by INTERHEART investigators and developed in the following paper: https://academic.oup.com/eurheartj/article/32/5/581/426790. The score consolidates multiple established risk factors for heart disease in addition to physical activity and diet, including psychosocial stress, lipids, smoking status, diabetes etc. Higher scores indicate greater predicted risk of heart attack and lower scores indicate lower risk of heart attack. The score ranges from 0 to 32. A one point increase in the score is associated with a 12% increased risk of having a heart attack.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Pare, MSc,MD,FRCPC, Principal Investigator — Hamilton Health Sciences, McMaster University
Locations (1):
- Hamilton Health Sciences (Juravinski Hospital, General Hospital, MUMC), Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Informed Consent Form (2018-02-24): https://cdn.clinicaltrials.gov/large-docs/83/NCT03583983/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2019-02-05): https://cdn.clinicaltrials.gov/large-docs/83/NCT03583983/Prot_SAP_002.pdf